CLINICAL TRIAL: NCT00137098
Title: Influence of Coffee on Heart Rate Variability Post Myocardial Infarction
Brief Title: Coronary Care Caffeine: Influence of Coffee on Heart Rate Post Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: The Royal Bournemouth Hospital (Other)
Other Study IDs: BDEC Caffeine
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Caffeine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Caffeine

SUMMARY:
Sudden cardiac death due to a heart rhythm disturbance after a heart attack (myocardial infarction) is a common cause of death. It is well documented that sudden cardiac death after a myocardial infarct (MI) is associated with low or poor heart rate variability (HRV). HRV is a measure of beat-to-beat changes in heart rate, with a greater variation associated with a "healthier" heart. The effect of caffeine on HRV in patients at high risk for sudden cardiac death is unknown. We, the investigators at the Royal Bournemouth Hospital, aim to study the effect of coffee or tea on HRV after MI.

DETAILED DESCRIPTION:
120 post MI patients on CCU will be studied during the first week of admission. Patients will be categorised using the following criteria: Infarct size and site; PMH; Co-morbidities; Drugs; Regular caffeine ingestion.

Patients will be randomised to receive either caffeinated or de-caffeinated coffee or tea during admission. HRV will be assessed by non-invasive Holter-monitoring on the fifth day. Salivary caffeine concentration will be assessed concurrently to assess compliance.

ELIGIBILITY:
Inclusion Criteria:

* ST-segment elevation (trans-mural) MI; sinus rhythm.
* Age < 80 years.

Exclusion Criteria:

* Cardiogenic shock
* Nothing by Mouth (NBM)
* Caffeine intolerance
* Atrial fibrillation, temporary or permanent pacing
* Complete heart block, bundle branch block, severe left ventricular impairment, non-ST segment MI/acute coronary syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of either gender, over 18 and under 80 years of age, admitted to the Coronary Care Unit following myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-09; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Richardson, Dr, Principal Investigator — Royal Bournemouth Hospital
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom